CLINICAL TRIAL: NCT06232343
Title: Effects of Parachute Resistance Training on Strength, Fatigue and Gait Parameters in Young Athletes
Brief Title: Effects of Parachute Resistance Training in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0760
Record Dates: First submitted 2023-12-26; First posted 2024-01-30 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Children, Only
Keywords: Gait; Resistance training; Speed; Strength

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This group followed a resisted training programmed with a parachute
  Interventions: Other: Parachute Resistance Training
- Controlled (Other): This group perform sprinters with no external resistance training
  Interventions: Other: Sprinters

INTERVENTIONS:
Other: Parachute Resistance Training — The training programmed duration is of four weeks.The groups will follow the training programmed three times a week. The daily schedule (training group) included four repetitions of maximum intensity 30 m & 50 m dashes (4 × 30 m, 4 × 50 m). The duration of recovery time between the 30 m & 50 m runs will be 4 and 6 minutes respectively. Between the last 30 m dash and the first 50 m dash, a 10-minute recovery will be applied. Moreover, sprint speed training should not exceed 400-500 meters in total . To this end, the training programmed of the present study consisted of 4x30m and 4x50m runs, at a frequency of 3 times a week.
  Arms: Experimental
Other: Sprinters — control group perform sprinters without any external resistance training for four weeks.
  Arms: Controlled

SUMMARY:
Muscular power may protect against cardiovascular disease independently of cardiorespiratory fitness. Resistance training is a useful training technique to boost running speed while enhancing other aspect of an athlete's physical condition. Resistance training is also consisting of weight training. Weight training emphasis on health exercise program. Improvements in muscular strength, power, running speed, kicking velocity, endurance, dynamic balance, flexibility, and general motor function have been observed in youth who have participated in resistance training between the ages of 8 to 14 years. These improvements strengthen young athletes' immunity to common sports ailments It will be Randomized Controlled trial in which convenient sampling technique will be used. Two groups will be formed in which participants will be divided by lottery method. Group A in which will be treated By Parachute resistance training and the other group will perform sprinters. Fatigue Assessment Scale and Strength 1RM tool will be used. The result after statistical analysis will either show this intervention is effective or not. Results will be analyzed on SPSS

DETAILED DESCRIPTION:
The study plan consisted of three parts, a) initial evaluation testing b) implementation of a 4-week intervention training programme c) evaluation retesting.

The resisted sprint training method will be adopted. To achieve resistance, a parachute will be used. The rate of applied resistance should be such that no alteration of the running technique would be observed. Any running velocity decrease 10% compared to un-resisted running indicates that the applied resistance load is too high and will have adverse effects on the sprinting technique.

The subjects will be divided randomly into two groups (Ν = 21each). Both groups will follow the same training programmed. The first group followed a resisted training programmed with a parachute (resisted group-RG), while the other group used no external resistance (un-resisted group-UG).control group perform sprinters. The training programmed will have duration of four weeks and will be implemented in the same facility in which the evaluation procedures will be held. The preparation/warm-up protocol throughout the training programmed will be the same with the protocol that was implemented during the testing procedures. The groups will follow the training programmed three times a week. The daily schedule (training group) included four repetitions of maximum intensity 30 m & 50 m dashes (4 × 30 m, 4 × 50 m). The duration of recovery time between the 30 m & 50 m runs will be 4 and 6 minutes respectively. Between the last 30 m dash and the first 50 m dash, a 10-minute recovery will be applied. With regard to the frequency and volume of the intervention programmed, sprint - speed training is characterized by maximum intensity stimuli to be repeated 2-4 times a week. Moreover, sprint - speed training should not exceed 400-500 meters in total . To this end, the training programmed of the present study consisted of 4x30m and 4x50m runs, at a frequency of 3 times a week. (Total volume = 120 m + 200 m = 320 m). The duration of the recovery time will be 4 and 6 minutes for the 30 m and 50 m runs respectively, and 10 minutes between each set. 4-minutes of recovery time is adequate for the body to reach full recovery. A recovery time longer than 12 minutes between repetitions in total results in inactivation of the central nervous system

ELIGIBILITY:
Inclusion Criteria:

* Age 08-14 years
* Athletic Participants will be included
* Both Gender Boys and Girls will be included

Exclusion Criteria:

* Participants with any musculoskeletal, neurological, cardiovascular, or respiratory disablements
* Those who were unable to complete follow-up tests.
* Participants with leg length discrepancy.
* Participants Previous surgery
* Participants are not currently using or ever used supplements that can effect muscles

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Fatigue | 4 weeks
  The Fatigue Assessment Scale (FAS) is a unidimensional fatigue scale to rate how a person usually feels that is scored using a 5-point Likert scale from 1 (never) to 5 (always). It consists of 10 items, 9 of which were derived from four useful fatigue scales, namely the Checklist Individual Strength (CIS), the Emotional Exhaustion subscale from the Dutch version of the Maslach Burnout Inventory, the Energy and Fatigue subscale from the World Health Organization Quality of Life assessment instrument, and the Fatigue Scale. The satisfactory reliability and content validity of FAS were confirmed. Moreover, this scale is short and easy to use. 10-22 no fatigue, 22-34 mild fatigue, 35-50 severe
Strength 1RM | 4 weeks
  The one-repetition maximum (1RM) is the heaviest weight that can be lifted just once while using proper form. There are a number of benefits of the 1RM test over traditional laboratory testing. The 1 repetition maximum test more accurately reflects the dynamic muscle actions that are most typically utilized in resistance training and of natural movement in most activities of sport and daily life since eccentric actions are usually paired with concentric actions. Strength in compound movements can be evaluated with the 1RM test. The "gold standard" of dynamic strength tests, according to many studies. One study conducted in the year 2020 found that ICCs might be anywhere from 0.64 to 0.99 (median ICC = 0.97), with the vast majority (92%) having values below 0.90 and the vast majority (97%) having values below 0.80. CVs were observed between 5% and 12.1 % (median CV = 4.2 %)
Gait parameters | 4 weeks
  1. Cadence (no. of step/time)
  2. Stride length (cm) distance of heel of right to heel of right
  3. Step length (cm) initial contact of one foot to initial contact of opposite foot
  4. Step width (cm) distance between two heels Speed (m/sec) distance/ time

CONTACTS AND LOCATIONS:
Overall Officials: Umme Ammara, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walters BK, Read CR, Estes AR. The effects of resistance training, overtraining, and early specialization on youth athlete injury and development. J Sports Med Phys Fitness. 2018 Sep;58(9):1339-1348. doi: 10.23736/S0022-4707.17.07409-6. Epub 2017 Jun 8. PMID 28597618
- [Background] Zwolski C, Quatman-Yates C, Paterno MV. Resistance Training in Youth: Laying the Foundation for Injury Prevention and Physical Literacy. Sports Health. 2017 Sep/Oct;9(5):436-443. doi: 10.1177/1941738117704153. Epub 2017 Apr 27. PMID 28447880